CLINICAL TRIAL: NCT00961168
Title: Prospective Study on the Effects of Artificial Breathing Patterns on Work of Breathing in Patients With Acute Lung Injury.
Brief Title: Work of Breathing and Mechanical Ventilation in Acute Lung Injury
Acronym: WOBALI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Budgetary restrictions
Sponsor: University of California, San Francisco (Other)
Responsible Party: Mitchell Cohen, MD, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: WOBARDS
Record Dates: First submitted 2009-08-16; First posted 2009-08-18 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Acute Lung Injury
Keywords: Mechanical Ventilation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lung-Protective Ventilation (Experimental): Lung-Protective Ventilation comparing volume vs. pressure control
  Interventions: Other: Volume Control Ventilation; Other: Pressure Control Ventilation

INTERVENTIONS:
Other: Volume Control Ventilation — Mechanical ventilation at a constant tidal volume of 6 mL/kg.
  Other Names: Volume Assist/Control
Other: Pressure Control Ventilation — Mechanical ventilation at a constant airway pressure of 25-30 cm H2O
  Other Names: Pressure Assist/Control

SUMMARY:
The primary goal of this study is to measure changes in biological markers of inflammation in critically-ill patients with acute lung injury (ALI) or acute respiratory distress syndrome (ARDS) while they are treated with different styles of lung-protective, artificial breathing assistance.

Secondary goals are to measure the breathing effort of patients using different artificial breathing patterns from the breathing machine.

The primary hypothesis is that volume-targeted artificial patterns will produce less inflammation. The secondary hypothesis is that volume-targeted artificial patterns will increase breathing effort compared to pressure-targeted artificial patterns.

DETAILED DESCRIPTION:
Ventilator-induced lung injury contributes to the progression of ALI/ARDS,1 and is thought to occur partly from the unequal distribution of a super-normal tidal volume to normal areas of the lung.2 Alveolar overdistension causes alveolar-capillary membrane damage,3 increased-permeability pulmonary edema4 and hyaline membrane formation.5 Therefore, it is recommended that tidal volume should be reduced to 6-7 mL/kg, and that the peak alveolar pressure, or the end-inspiratory plateau pressure (PPLAT), should be limited to < 30 cm H2O.6 The National Heart Lung and Blood Institute's ARDS Network demonstrated a 22% reduction in mortality using a "lung-protective" (low tidal volume) ventilation strategy in patients with ALI/ARDS.7 High tidal volume ventilation causes a rapid and substantial increase plasma levels of proinflammatory mediators which decrease in response to lung protective ventilation.8,9 A consequence of lung-protective ventilation is dyspnea and increased work of breathing.10 Our recent study11 on work of breathing during lung-protective ventilation found that inspiratory pleural pressure changes were extraordinarily high, averaging 15-17 cm H2O. Whereas tidal volume was well controlled during volume ventilation, in contrast, it exceeded target levels in 40% of patients during pressure control ventilation.

High tidal volume-high negative pressure ventilation causes acute lung injury in animal models.12,13 Thus ventilator-induced lung injury results from excessive stress across lung tissue created by high transpulmonary (airway-pleural).pressure.14 This suggests the possibility that despite pressure control ventilation being set with a low positive airway pressure, "occult" high tidal volume-high transpulmonary pressure ventilation still may occur.11 However, during spontaneous breathing diaphragmatic contractions cause ventilation to be distributed preferentially to dorsal:caudal aspects of the lungs.15 Therefore, high transpulmonary pressures created by large negative swings in pleural pressure theoretically may not cause regional lung over-distension and ventilator-induced lung injury if tidal ventilation is preferentially distributed to dorsocaudal lung regions. However, a study16 examining the effects of diaphragmatic breathing during Pressure Control Ventilation found that dorsocaudal distribution of tidal volume was not necessarily improved compared to passive ventilation, as the amount of tidal ventilation distributed to areas of high ventilation/perfusion was unaltered. Regardless, during a recent conference on respiratory controversies in the critical care setting, it was noted that the effects of ventilator modes such as volume control, pressure control and airway pressure-release ventilation on proinflammatory cytokine expression during lung-protective ventilation has not been studied in humans.17 Thus it is unknown whether or not differences in transpulmonary pressure and tidal volume between these modes has a direct impact on lung inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Both medical and surgical patients undergoing mechanical ventilatory support who meet criteria for Acute Lung Injury (ALI) or Acute Respiratory Distress Syndrome (ARDS) as defined by the European-American Consensus Conference,
* Mechanical ventilation via an endotracheal or tracheotomy tube,
* PaO2/FiO2 < 300 mmHg with bilateral infiltrates on chest radiogram,
* Clinical management with lung protective ventilation (Tidal volume < 8 mL/kg).

Exclusion Criteria:

* Patients receiving "comfort care",
* High cervical spinal cord injury or other neuromuscular disease,
* Prisoners,
* Pregnancy,
* Less than 18 years of age,
* Facial fractures and coagulopathies,
* Patients placed on psychiatric hold.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
proinflammatory cytokine expression in plasma | 2 hours

SECONDARY OUTCOMES:
work of breathing | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cohen, MD, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Background] 1. Dreyfus D, Sauman G. Ventilation induced injury. In: Principles and Practice of Mechanical Ventilation. Tobin M J. Editor. New York: McGraw Hill Publishers; 1994: 793-811.
- [Background] Hickling KG. Ventilatory management of ARDS: can it affect the outcome? Intensive Care Med. 1990;16(4):219-26. doi: 10.1007/BF01705155. PMID 2193041
- [Background] Fu Z, Costello ML, Tsukimoto K, Prediletto R, Elliott AR, Mathieu-Costello O, West JB. High lung volume increases stress failure in pulmonary capillaries. J Appl Physiol (1985). 1992 Jul;73(1):123-33. doi: 10.1152/jappl.1992.73.1.123. PMID 1506359
- [Background] Carlton DP, Cummings JJ, Scheerer RG, Poulain FR, Bland RD. Lung overexpansion increases pulmonary microvascular protein permeability in young lambs. J Appl Physiol (1985). 1990 Aug;69(2):577-83. doi: 10.1152/jappl.1990.69.2.577. PMID 2228868
- [Background] Lachmann B, Jonson B, Lindroth M, Robertson B. Modes of artificial ventilation in severe respiratory distress syndrome. Lung function and morphology in rabbits after wash-out of alveolar surfactant. Crit Care Med. 1982 Nov;10(11):724-32. doi: 10.1097/00003246-198211000-00005. No abstract available. PMID 6754260
- [Background] 6. Tuxen DV. Permisive hypercapnia. In: Principles and Practice of Mechanical Ventilation. Tobin M J. Editor. New York: McGraw Hill Publishers; 1994: 371-392.
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Ranieri VM, Suter PM, Tortorella C, De Tullio R, Dayer JM, Brienza A, Bruno F, Slutsky AS. Effect of mechanical ventilation on inflammatory mediators in patients with acute respiratory distress syndrome: a randomized controlled trial. JAMA. 1999 Jul 7;282(1):54-61. doi: 10.1001/jama.282.1.54. PMID 10404912
- [Background] Stuber F, Wrigge H, Schroeder S, Wetegrove S, Zinserling J, Hoeft A, Putensen C. Kinetic and reversibility of mechanical ventilation-associated pulmonary and systemic inflammatory response in patients with acute lung injury. Intensive Care Med. 2002 Jul;28(7):834-41. doi: 10.1007/s00134-002-1321-7. Epub 2002 Jun 15. PMID 12122519
- [Background] Tuxen DV. Permissive hypercapnic ventilation. Am J Respir Crit Care Med. 1994 Sep;150(3):870-4. doi: 10.1164/ajrccm.150.3.8087364. No abstract available.
- [Background] Kallet RH, Campbell AR, Dicker RA, Katz JA, Mackersie RC. Work of breathing during lung-protective ventilation in patients with acute lung injury and acute respiratory distress syndrome: a comparison between volume and pressure-regulated breathing modes. Respir Care. 2005 Dec;50(12):1623-31. PMID 16318643
- [Background] Dreyfuss D, Soler P, Basset G, Saumon G. High inflation pressure pulmonary edema. Respective effects of high airway pressure, high tidal volume, and positive end-expiratory pressure. Am Rev Respir Dis. 1988 May;137(5):1159-64. doi: 10.1164/ajrccm/137.5.1159. PMID 3057957
- [Background] Mascheroni D, Kolobow T, Fumagalli R, Moretti MP, Chen V, Buckhold D. Acute respiratory failure following pharmacologically induced hyperventilation: an experimental animal study. Intensive Care Med. 1988;15(1):8-14. doi: 10.1007/BF00255628. PMID 3230208
- [Background] Gattinoni L, Pesenti A. The concept of "baby lung". Intensive Care Med. 2005 Jun;31(6):776-84. doi: 10.1007/s00134-005-2627-z. Epub 2005 Apr 6. PMID 15812622
- [Background] Froese AB, Bryan AC. Effects of anesthesia and paralysis on diaphragmatic mechanics in man. Anesthesiology. 1974 Sep;41(3):242-55. doi: 10.1097/00000542-197409000-00006. No abstract available. PMID 4604401
- [Background] Myers TR, MacIntyre NR. Respiratory controversies in the critical care setting. Does airway pressure release ventilation offer important new advantages in mechanical ventilator support? Respir Care. 2007 Apr;52(4):452-8; discussion 458-60. PMID 17417979